CLINICAL TRIAL: NCT00640757
Title: Methionine-Restriction Diet (MRD) in Obese Adults With Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Orentreich Foundation for the Advancement of Science, Inc. (Other)
Responsible Party: Principal Investigator, Frank Greenway, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 26009
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Metabolic Syndrome
Keywords: Methionine; Metabolic syndrome; Glucose Metabolism; Amino acid; Insulin clamp
MeSH Terms: conditions — Metabolic Syndrome | interventions — Methionine; Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Methionine 1 (Active Comparator): Methionine deficient diet
  Interventions: Dietary Supplement: Methionine deficient diet
- Placebo 2 (Placebo Comparator): Placebo comparator methionine complete diet
  Interventions: Dietary Supplement: Methionine sufficient diet

INTERVENTIONS:
Dietary Supplement: Methionine deficient diet — Hominex with a low protein diet
  Other Names: Hominex; Methionine
  Arms: Low Methionine 1
Dietary Supplement: Methionine sufficient diet — Hominex, low protein diet and methionine capsules
  Other Names: Hominex; Methionine capsules; Low protein diet
  Arms: Placebo 2

SUMMARY:
The purpose of this study is to determine if limiting dietary methionine (MET), one of the 10 essential amino acids (which make up proteins), causes weight loss and/or improves glucose metabolism.

DETAILED DESCRIPTION:
Methionine deficient diets have been shown to increase metabolic rate, decrease weight and extend lifespan in rodents. A methionine deficient diet has been tested for 17 weeks in humans without adverse events and with an average weight loss of 8 kg. This study will test the ability of a low methionine diet to cause weight loss and improve the metabolic syndrome. The metabolic syndrome is driven by insulin resistance which is associated with abdominal fat, so this study hopes to reduce visceral fat, body weight and improve insulin resistance.

Twenty-four healthy males or females 21 to 60 years of age, inclusive with a stable weight and a waist circumference >40" in men and >35" in women will participate in this study. Subjects will need at least two of the following: 1) HDL cholesterol < 40 mg/dL in men or < 50 mg/dl in women; 2) triglycerides > 150 mg/dL, 3) blood pressure >130/85 mmHg; 4) fasting glucose 110-125 mg/dL. Subjects who have diabetes, a history of heart attack, stroke, have had cancer in the last five years or take chronic medication for a significant illness will be excluded.

Subjects will have a medical history, physical examination, chemistry panel, complete blood count (CBC), electrocardiogram, DEXA, abdominal CT scan to quantitate visceral fat, and blood will be sent to Orentreich for glucose, insulin, C-peptide, lipid profile with particle size, free fatty acids, adiponectin, leptin, high-sensitivity C-reactive protein, and insulin-like growth factor-1. Subjects will also undergo a hyperinsulinemic, euglycemic clamp to quantitate insulin resistance during an 18 hr inpatient stay, and will spend 24 hours in the metabolic chamber to measure metabolic rate. Subjects will then be placed on a diet of Hominex-2, a drink that will give them their protein in an amount based on their body weight, and they will see a dietitian who will give them a list of food they can eat consisting mainly of fruits, vegetables and a small amount of grains. Calories will not be restricted and subjects will receive a choline supplement of 500 mg/d. Subjects will be randomized to receive capsules containing methionine or placebo based on their body weight. The two groups will be on 2mg/kg/d or 23 mg/kg/d of methionine.

Participants will return to PBRC every 2 weeks throughout the 16-week diet period to meet with the dietician, have weight and vital signs recorded, and have fasting blood drawn every 4 weeks to be sent to Orentreich for compliance measures.

The physical exam, multi-slice CT scan, DEXA, inpatient admission for euglycemic hyperinsulinemic clamp, metabolic chamber stay, and the blood testing obtained at screening and baseline will be repeated at the completion of the 16 week diet period.

There are no known risks to the low methionine diet, but some people may have gastrointestinal upsets when they change their diet. The risk of the CT scan is exposure to x-radiation equivalent to a front and side view chest x-ray. The risk of the DEXA is the exposure to x-irradiation equivalent to spending 12 hours in the sunshine. There are no risks to staying in the metabolic chamber. The hyperinsulinemic, euglycemic clamp could cause low blood sugar. This will be avoided by frequent monitoring of blood sugar, and if the low blood sugar were to occur, the test would be stopped and sugar given through the intravenous line. The testing of blood involves the discomfort of a needle going into an arm vein, bruising and rarely fainting or infection. These risks will be minimized by trained technicians using sterile needles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21 to 60, inclusive
* Waist greater than 40 inches for men and 35 inches for women
* Weight has been stable for at least 6 months (no more than 5 pounds gained or lost)
* For women of childbearing potential: subject must be willing to use acceptable form of contraception (pill, condom, diaphragm etc.)
* At least 2 of the following:

HDL cholesterol

* Men < 40 mg/dL
* Women < 50 mg/dL Triglycerides ≥150 mg/dL Blood pressure ≥130/≥ 85 mmHg Fasting glucose ≥110-125 mg/dL

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* History of heart attack or stroke
* Pregnant or breastfeeding or planning to become pregnant during the study
* Cancer (other than non-melanoma skin) within the last 5 years
* Significant illness requiring medication
* Inability to read and follow directions in English
* Donated blood in the last 2 months.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | Every 2 weeks

SECONDARY OUTCOMES:
Improve glucose metabolism | Baseline and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Gettys, Ph.D., Principal Investigator — Pennington Biomedical Research Center

REFERENCES:
- [Derived] Plaisance EP, Greenway FL, Boudreau A, Hill KL, Johnson WD, Krajcik RA, Perrone CE, Orentreich N, Cefalu WT, Gettys TW. Dietary methionine restriction increases fat oxidation in obese adults with metabolic syndrome. J Clin Endocrinol Metab. 2011 May;96(5):E836-40. doi: 10.1210/jc.2010-2493. Epub 2011 Feb 23. PMID 21346062